CLINICAL TRIAL: NCT04970030
Title: Comparison Between Mechanical Intracanal (ML) Lithotripsy and Electrohydraulic Intracolangioscopic (EHL) Lithotripsy in the Treatment of Difficult Main Biliary Tract Lithiasis
Acronym: ML_vs_EHL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 397-2021-SPER-AUSLBO
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Gallstone; Lithiasis
Keywords: Gallstone, Lithiasis, ML lithotripsy, EHL lithotripsy
MeSH Terms: conditions — Gallstones; Lithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mechanical intracanal (ML) lithotripsy (Active Comparator): TTS mechanical lithotripter
  Interventions: Procedure: ML lithotripsy
- electrohydraulic intracolangioscopic (EHL) lithotripsy (Experimental): electrohydraulic lithotripsy with Autolith probe
  Interventions: Procedure: EHL lithotripsy

INTERVENTIONS:
Procedure: ML lithotripsy — we will proceed under fluoroscopic vision with TTS mechanical lithotripter (Trapezoid, RX Wireguided Retrieval Basket, Boston Scientific) with mechanical fragmentation of the stone and subsequent complete cleaning of the biliary tract using the fluoroscopic technique.
  Arms: mechanical intracanal (ML) lithotripsy
Procedure: EHL lithotripsy — after administration of IV antibiotic therapy, we will proceed to cholangioscopy with SpyGlass ™ DS (Boston Scientific Corporation, USA), treatment of difficult biliary lithiasis with electrohydraulic lithotripsy with Autolith probe (Northgate Technologies Inc USA) and subsequent complete cleaning of the biliary tract using the fluoroscopic technique
  Arms: electrohydraulic intracolangioscopic (EHL) lithotripsy

SUMMARY:
Difficult gallstones are found in about 10-15% of endoscopic retrograde cholangiopancreaticography (ERCP) performed for choledocholithiasis. There are several options for the treatment of difficult biliary lithiasis including mechanical lithotripsy and peroral cholangioscopy with electrohydraulic lithotripsy.

The primary purpose of this study is to compare the effectiveness of treating difficult biliary lithiasis with ML and with EHL. The effectiveness is defined by the complete cleanliness of the biliary tract in a single endoscopic session

DETAILED DESCRIPTION:
Difficult gallstones are found in about 10-15% of endoscopic retrograde cholangiopancreaticography (ERCP) performed for choledocholithiasis. There are several options for the treatment of difficult biliary lithiasis including mechanical lithotripsy and peroral cholangioscopy with electrohydraulic lithotripsy.

The primary purpose of this study is to compare the effectiveness of treating difficult biliary lithiasis with ML and with EHL. The effectiveness is defined by the complete cleanliness of the biliary tract in a single endoscopic session.

The secondary objectives of the study are as follows:

* Within 30 days of the procedure, the effective clearance of the biliary tract will be assessed with CholangioRM (or EUS where MRI is contraindicated). If residual choledocholithiasis is present, patients will be considered as late failures.
* Comparison of the safety of the treatments under study, defined by the incidence of adverse events during the procedure (e.g. perforation, hemobilia) and in the observation period after the procedure (e.g. cholangitis, pancreatitis, bleeding).

Patients that can be enrolled:

All patients with "difficult" biliary tract lithiasis that could not be treated by standard techniques, such as balloon and/or basket catheter under fluoroscopic vision.

Patients cannot be enrolled:

* if they have a surgically-altered gastrointestinal anatomy
* if they have any evidence of biliopancreatic malignancy
* if they are under 18 years of age
* if they are in a state of pregnancy or are breastfeeding
* if it's impossible to obtain informed consent

If, while performing ERCP for choledocholithiasis, stones are found that cannot be removed using standard treatment, they will be treated by assigning these patients to either the treatment group with ML under fluoroscopic vision or to the EHL treatment group.

Patients will be assigned using a randomization method in blocks with a ratio of 1:1 for each patient enrolled.

Subjects will undergo ERCP, either under general anesthesia, or under observation by an anesthesiologist, and depending on which group they have been assigned to, will be treated with:

* EHL: after administration of IV antibiotic therapy, we will proceed to cholangioscopy with SpyGlass ™ DS (Boston Scientific Corporation, USA), treatment of difficult biliary lithiasis with electrohydraulic lithotripsy with Autolith probe (Northgate Technologies Inc USA) and subsequent complete cleaning of the biliary tract using the fluoroscopic technique.
* ML: we will proceed under fluoroscopic vision with TTS mechanical lithotripter (Trapezoid, RX Wireguided Retrieval Basket, Boston Scientific) with mechanical fragmentation of the stone and subsequent complete cleaning of the biliary tract using the fluoroscopic technique.

During each procedure, the following will be recorded:

* the execution time from the insertion of the cholangioscope or lithotripter inside the biliary tract until the complete cleaning of the biliary tract is finished.
* the occurrence of possible adverse events related to the procedures and/or anesthetic issues.
* any failure of a technique and / or the need to switch a patient to the other treatment group.

At least 50 patients eligible for the study will be required.

ELIGIBILITY:
Inclusion Criteria:

- All patients with "difficult" biliary tract lithiasis that could not be treated by standard techniques, such as balloon and/or basket catheter under fluoroscopic vision.

Exclusion Criteria:

* surgically-altered gastrointestinal anatomy
* any evidence of biliopancreatic malignancy
* patients under 18 years of age
* patients in a state of pregnancy or are breastfeeding
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
ML - EHL comparison | 1 day
  The primary purpose of this study is to compare the effectiveness of treating difficult biliary lithiasis with ML and with EHL. The effectiveness is defined by the complete cleanliness of the biliary tract in a single endoscopic session

SECONDARY OUTCOMES:
effective clearance of the biliary tract | 30 days
  Within 30 days of the procedure, the effective clearance of the biliary tract will be assessed with CholangioRM (or EUS where MRI is contraindicated). If residual choledocholithiasis is present, patients will be considered as late failures.
Comparison of the safety of the treatments under study | 30 days
  Comparison of the safety of the treatments under study, defined by the incidence of adverse events during the procedure (e.g. perforation, hemobilia) and in the observation period after the procedure (e.g. cholangitis, pancreatitis, bleeding).

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No